CLINICAL TRIAL: NCT01465854
Title: French Biological Observatory on Lung Cancer in Never Smokers
Acronym: BioCAST
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Other Study IDs: IFCT-1002 BioCAST
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
Keywords: lung cancer; smoking; molecular epidemiology; genetic polymorphism; risk factors; never smokers; histologically/cytologically confirmed; IFCT
MeSH Terms: conditions — Lung Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plama, white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LCINS: Never smokers with newly diagnosed lung cancer

SUMMARY:
Lung cancer in non-smokers (LCINS) is an increasing public health problem. The BioCAST (IFCT-1002) study, promoted by Intergroupe Francophone de Cancérologie Thoracique (IFCT), focuses on this entity. It is a national, multicentric, prospective epidemiological study. Main objective is to describe the clinical and molecular epidemiology of LCINS in a large French cohort composed by cases newly diagnosed in participating centres (around to 1000 patients expected). The clinical component of the study is based on collecting data directly from the patient through a standardized questionnaire during a telephone interview with a health professional. The biologic component includes a blood sample collection. A large genomic-wide association study and an epigenetic study are also planned. BioCAST hopes to provide concrete answers to clinicians and patients questions about this new and frequent entity.

DETAILED DESCRIPTION:
According to WHO, 25% of lung cancer worldwide occurs in lifelong never smokers. Lung cancer in never smokers (LCINS) shows many clinical, epidemiological, molecular and genomic differences comparing to tobacco-related neoplasm. So, it is now considered as a separate entity. LCINS particularly occurs in women and Asian. They are mainly adenocarcinoma. Known risk factors are occupational exposure, environmental tobacco smoking, familial history of cancer, personal medical history of lung disease or environmental causes. LCINS carries more frequently molecular abnormalities leading to efficacy of targeted therapies (EGFR mutation, EML4-ALK inversion, less frequent mutations of KRAS ...). However, most data come from retrospectives studies, subgroups analysis and/or from Asian cohort even though it is a disease with a significant geographic variability. Finally, few studies focus on correlations between risk factors and molecular or genomic abnormalities.

For these reasons and considering that LCINS is an increasing public health problem, IFCT (Intergroupe Francophone de Cancérologie Thoracique) states to promote the BioCAST study (IFCT-1002). It is a national, multicentric, prospective epidemiological study. Main objective is to describe the clinical and molecular epidemiology of LCINS in a French population composed by all cases newly diagnosed in participating centres (500 to 1500 patients expected). BioCAST include a clinical and a biological part. The clinical component is based on collecting data directly from the patient through a standardized questionnaire during a telephone interview with a health professional. The biologic component includes a blood sample collection. A large genomic wide association study and an epigenetic study (including micro RNA study) are also planned. Other objectives are looking for correlations between clinical factors and molecular abnormalities; and looking for new oncogene in this specific population.

BioCAST hopes to provide concrete answers to clinicians and patients about this new and frequent entity.

ELIGIBILITY:
Inclusion Criteria:

* never smokers (i.e. who has smoked less than 100 cigarettes per lifetime)
* at least 18 years of age
* newly diagnosed lung cancer
* patient having access to a telephone
* french-speaking patient or patient who could be easily helped in his mother tongue during a phone interview
* signed informed consent

Exclusion Criteria:

* smokers
* chemotherapy already initiated at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Never smokers with newly diagnosed lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of EGFR mutations in never smokers with newly diagnosed non-small-cell lung cancer (NSCLC) | November 2011 to January 2013

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien COURAUD, MD, Principal Investigator — Hospices Civils de Lyon, CH Lyon Sud, FRANCE
Locations (82):
- France (82):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - CHD Castelluccio, Ajaccio
  - Clinique Claude Bernard, Albi
  - CHU d'Angers, Angers
  - CHI Annemasse-Bonneville, Annemasse
  - CH Annonay, Annonay
  - Hôpital Privé d'Antony, Antony
  - CHIC, Aulnay-sous-Bois
  - CH de la Côte Basque, Bayonne
  - CHU Besançon, Besançon
  - Hôpital Ambroise Paré - Pneumologie, Boulogne
  - Hôpital Fleyriat, Bourg-en-Bresse
  - CH Jacques-Cœur - Pneumologie, Bourges
  - CH Pierre Oudot, Bourgoin
  - HCL Hôpital Louis Pradel, Bron
  - Centre François Baclesse, Caen
  - CHU Côte de Nâcre, Caen
  - CH Cahors, Cahors
  - CH de Cannes, Cannes
  - CH Chambery, Chambéry
  - CH de Chartres Hôpital Louis Pasteur, Chartres
  - CH de Chauny, Chauny
  - Centre Médical Nicolas de Pontoux, Châlon-sur-Saône
  - CH de Châlons-en-Champagne, Châlons-en-Champagne
  - Hôpital de Cholet - Pneumologie, Cholet
  - HIA Percy - Pneumologie, Clamart
  - Hôpitral Gabriel Montpied - Pneumologie, Clermont-Ferrand
  - Hôpital Pasteur, Colmar
  - CH Compiègne - Pneumologie, Compiègne
  - CHI Créteil, Créteil
  - CH de Dax, Dax
  - Cabinet privé, Dijon
  - Centre d'Oncologie du Parc, Dijon
  - Centre Georges François Leclerc, Dijon
  - CHU Hôpital du Bocage, Dijon
  - CHRU Grenoble, Grenoble
  - CH Région Saint-Omer, Helfaut
  - CH Lagny-sur-Marne, Lagny-sur-Marne
  - CH de Versailles, Le Chesnay
  - CH du Mans, Le Mans
  - Centre Oscar Lambret, Lille
  - Hôpital Calmette, Lille
  - CH de Longjumeau, Longjumeau
  - CH Lyon Sud - Pneumologie, Lyon
  - CH Saint Joseph Saint Luc, Lyon
  - Clinique Mutualiste Eugène André, Lyon
  - HIA Desgenettes, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Ambroise Paré, Marseille
  - Hôpital Nord - Oncologie Multidisciplinaire & Innovations Thérapeutiques, Marseille
  - Polyclinique du Parc, Maubeuge
  - CH de Macon, Mâcon
  - CHR Metz Thionville, Metz
  - CH de Mont-De-Marsan, Mont-de-Marsan
  - CH Montélimar, Montélimar
  - CH de Mulhouse, Mulhouse
  - CHU Nancy, Nancy
  - Hôpital Laënnec - CHU de Nantes, Nantes
  - CH Nevers, Nevers
  - Centre Antoine Lacassagne, Nice
  - CHR d'Orléans La Source, Orléans
  - GH Paris Saint-Joseph, Paris
  - Hôpital Bichat - Claude - Bernard, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Tenon, Paris
  - CH de Rambouillet, Rambouillet
  - Institut Jean Godinot, Reims
  - CHU Charles Nicolle, Rouen
  - CH de Saint-Brieuc, Saint-Brieuc
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHU Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpitaux du Léman - Pneumologie et Maladies Infectieuses, Thonon-les-Bains
  - Hôpital Font-Pré - Pneumologie, Toulon
  - Clinique Pasteur, Toulouse
  - Clinique Saint Jean du Languedoc, Toulouse
  - Hôpital Larrey - Pneumologie, Toulouse
  - CHU Tours - Pneumologie, Tours
  - CH Valence, Valence
  - CHI de la Haute-Saône - Pneumologie, Vesoul
  - Clinique Mutualiste Les Portes du Sud, Vénissieux
  - CH de Villefranche - Pneumologie, Villefranche

REFERENCES:
- [Result] Couraud S, Debieuvre D, Moreau L, Dumont P, Margery J, Quoix E, Duvert B, Cellerin L, Baize N, Taviot B, Coudurier M, Cadranel J, Missy P, Morin F, Mornex JF, Zalcman G, Souquet PJ; BioCAST/IFCT-1002 study investigators. No impact of passive smoke on the somatic profile of lung cancers in never-smokers. Eur Respir J. 2015 May;45(5):1415-25. doi: 10.1183/09031936.00097314. Epub 2015 Mar 5. PMID 25745045
- [Result] Couraud S, Souquet PJ, Paris C, Do P, Doubre H, Pichon E, Dixmier A, Monnet I, Etienne-Mastroianni B, Vincent M, Tredaniel J, Perrichon M, Foucher P, Coudert B, Moro-Sibilot D, Dansin E, Labonne S, Missy P, Morin F, Blanche H, Zalcman G; French Cooperative Intergroup IFCT. BioCAST/IFCT-1002: epidemiological and molecular features of lung cancer in never-smokers. Eur Respir J. 2015 May;45(5):1403-14. doi: 10.1183/09031936.00097214. Epub 2015 Feb 5. PMID 25657019
- [Result] Couraud S, Vaca-Paniagua F, Villar S, Oliver J, Schuster T, Blanche H, Girard N, Tredaniel J, Guilleminault L, Gervais R, Prim N, Vincent M, Margery J, Larive S, Foucher P, Duvert B, Vallee M, Le Calvez-Kelm F, McKay J, Missy P, Morin F, Zalcman G, Olivier M, Souquet PJ; BioCAST/IFCT-1002 investigators. Noninvasive diagnosis of actionable mutations by deep sequencing of circulating free DNA in lung cancer from never-smokers: a proof-of-concept study from BioCAST/IFCT-1002. Clin Cancer Res. 2014 Sep 1;20(17):4613-24. doi: 10.1158/1078-0432.CCR-13-3063. Epub 2014 Jul 10. PMID 25013125
- [Result] Couraud S, Labonne S, Missy P, Morin F, Tran Q, Deroy A, Milleron B, Blanche H, Zalcman G, Souquet PJ; les membres du Groupe de travail << non-fumeurs de l'IFCT >>. [Lung cancer in never smokers: a French national cohort (BioCAST/IFCT-1002)]. Rev Mal Respir. 2013 Sep;30(7):576-83. doi: 10.1016/j.rmr.2013.03.006. Epub 2013 May 18. French. PMID 24034464
- [Result] Fontaine-Delaruelle C, Mazieres J, Cadranel J, Mastroianni B, Dubos-Arvis C, Dumont P, Monnet I, Pichon E, Locatelli-Sanchez M, Dixmier A, Coudert B, Fraboulet S, Foucher P, Dansin E, Baize N, Vincent M, Missy P, Morin F, Moro-Sibilot D, Couraud S; IFCT10-02 BioCAST investigators. Somatic profile in lung cancers is associated to reproductive factors in never-smokers women: Results from the IFCT-1002 BioCAST study. Respir Med Res. 2020 Mar;77:58-66. doi: 10.1016/j.resmer.2020.01.003. Epub 2020 Jan 31. PMID 32416585
- [Result] Paris C, Do P, Mastroianni B, Dixmier A, Dumont P, Pichon E, Chouaid C, Coudert B, Foucher P, Fraboulet S, Locatelli-Sanchez M, Baize N, Dansin E, Moreau L, Vincent M, Missy P, Morin F, Moro-Sibilot D, Couraud S; BioCAST/IFCT-1002 study investigators; to the BioCAST/IFCT- 1002 study. Association between lung cancer somatic mutations and occupational exposure in never-smokers. Eur Respir J. 2017 Oct 26;50(4):1700716. doi: 10.1183/13993003.00716-2017. Print 2017 Oct. PMID 29074543
- See also: Official website — http://www.ifct.fr/